CLINICAL TRIAL: NCT06403709
Title: Phase II Study of Irinotecan Plus Trifluridine/Tipiracil (TAS-102) in Combination With Bevacizumab as a Third-Line or Beyond Therapy for Patients With Metastatic Colorectal Cancer (mCRC)
Brief Title: Irinotecan, TAS-102 Plus Bevacizumab as a Third-Line or Beyond Therapy in mCRC Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SH-2023005
Record Dates: First submitted 2024-04-01; First posted 2024-05-08 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Trifluridine; tipiracil; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irinotecan, TAS-102 plus Bevacizumab arm (Experimental): Patients received an intravenous infusion of irinotecan (150mg/m2 on day 1) plus bevacizumab (5 mg/kg on day 1) and an oral administration of TAS-102(30 mg/m2 given bid on days 1-5), repeated every 14 days.
  Interventions: Drug: Irinotecan, Trifluridine/tipiracil (TAS-102) plus Bevacizumab

INTERVENTIONS:
Drug: Irinotecan, Trifluridine/tipiracil (TAS-102) plus Bevacizumab — These patients received an intravenous infusion of irinotecan (150mg/m2 on day 1) plus bevacizumab (5 mg/kg on day 1) and an oral administration of TAS-102(30 mg/m2 given bid on days 1-5), repeated every 14 days.
  Other Names: Irinotecan+TAS-102+Bevacizumab

SUMMARY:
Currently, the approved third-line treatments for metastatic colorectal cancer (mCRC) include regorafenib, fruquintinib, and trifluridine/tipiracil(TAS-102). In recent years, several phase I/II studies evaluated the combination of TAS-102 and bevacizumab in mCRC patients who were refractory to standard therapies and showed promising antitumor efficacy and manageable toxicity. In this single-center phase II study, the investigators explored the efficacy and safety of irinotecan, TAS-102, plus bevacizumab in a third-line or beyond therapy for patients with mCRC.

DETAILED DESCRIPTION:
The mCRC patients who are refractory to standard therapies and need a third-line or beyond therapy are eligible. Patients who previously received irinotecan while progressing during maintenance therapy are also eligible.

These patients received an intravenous infusion of irinotecan (150mg/m2 on day 1) plus bevacizumab (5 mg/kg on day 1) and an oral administration of TAS-102(30 mg/m2 given bid on days 1-5), repeated every 14 days.

The primary endpoint was the objective response rate (ORR), and the secondary endpoints included progression-free survival (PFS), overall survival (OS), and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Colorectal adenocarcinoma confirmed histologically or histopathologically.
2. Patients were clinically diagnosed with metastatic colorectal cancer based on computed tomography (CT) scan and magnetic resonance imaging (MRI) according to AJCC 8th edition.
3. Patients must have received standard therapy for mCRC and is refractory or intolerant to those therapies.
4. Age ≥18 and ≤70.
5. ECOG physical status score is 0 or 1, and no obvious deterioration within 2 weeks prior to use on Day 1 of Cycle 1.
6. Appropriate organ function according to the following laboratory test values:

   1. Hemoglobin value ≥90g/L.
   2. White blood cell count ≥3.5*109/L.
   3. Absolute neutrophil count ≥1.5*109/L.
   4. Platelet count ≥100*109/L.
   5. Serum creatinine ≤ upper limit of normal (ULN) or creatinine clearance ≥60ml/min.
   6. Total serum bilirubin ≤1.5* upper normal limit (ULN).
   7. Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤2.5* upper limit of normal value (ULN).
7. Signed the informed consent.

Exclusion Criteria:

1. The pathological types were squamous carcinoma, neuroendocrine carcinoma, adenosquamous carcinoma, and other histological types except adenocarcinoma.
2. Patients who had shown hypersensitivity to Irinotecan and Trifluridine/tipiracil (TAS-102) or any other component of them. Patients who previously received irinotecan while disease progressed. However, patients who previously received irinotecan while progressing during maintenance therapy are eligible.
3. Known hypersensitivity to Bevacizumab or hypersensitivity to any other component of Bevacizumab.
4. Patients unable to swallow or lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication.
5. Patients had recurrent episodes of bleeding (risk of gastrointestinal bleeding) or received transfusions in the previous 2 weeks.
6. Major surgery in the previous 4 weeks. (Biopsy is excluded)
7. Previous or concurrent cancer diagnosed within 5 years prior to study inclusion, except for curatively treated in situ cervical cancer, non-melanoma skin cancer, basal cell carcinoma, benign prostate cancer, ductal carcinoma in situ, well-differentiated thyroid cancers and superficial bladder tumors: staged Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor with lamina propria invasion). Carcinomas that can be cured by adequate treatment are also excluded.
8. History of abdominal fistula, gastro-intestinal perforation, intestinal obstruction, chronic diarrhea or inflammatory bowel disease including Crohns disease and ulcerative colitis within 6 months prior to the first study treatment.
9. Patients with severe cardiac dysfunction, such as LVEF< 50%, CHF≥ grade 2, severe/unstable angina, history of stroke or transient ischemic attack or myocardial infarction in the previous 6 months.
10. Uncontrolled hypertension (systolic blood pressure >160 mmHg or diastolic pressure >100 mmHg despite treatment) and uncontrolled diabetes (fasting plasma glucose > 8.9 mmol/l).
11. Patients with a history of ventricular tachycardia, torsades de pointes, prolonged QTc, complete left bundle branch block or third-degree atrioventricular conduction block..
12. Patients with active hepatitis B, hepatitis C, syphilis or human immunodeficiency virus infection.
13. Arterial or venous thrombotic or embolic events such as deep vein thrombosis, and pulmonary embolism within 6 months of starting study treatment (catheter-related thrombosis is excluded).
14. Patients with active pulmonary tuberculosis were taking anti-tuberculosis treatment or have taken anti-tuberculosis treatment within 12 months of starting study treatment.
15. Patients with severe primary respiratory diseases, interstitial lung disease, or history of pneumonitis.
16. Patients with current active infections requiring anti-infection treatment within 2 weeks of starting study treatment.
17. Patients with a history of psychiatric drug abuse or a history of drug abuse.
18. Pregnant or lactating women.
19. Patients of childbearing potential are unwilling to practice contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 36 months
  The proportion of patients with a confirmed complete response or partial response using RECIST 1.1

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 36 months
  The time from the date of the first administration of this regimen to the date of first documented disease progression or death due to any cause
Overall Survival (OS) | 36 months
  The time from the initiation of the first dose of medication in a patient to death from any cause.
Safety and tolerability by incidence, severity and outcome of adverse events | 36 months
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Yongkun Sun, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Beijing Chaoyang Sanhuan Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No